CLINICAL TRIAL: NCT07189793
Title: Toripalimab With Sequential Intravesical Gemcitabine-Mitomycin C Versus Toripalimab Alone for the Treatment of BCG-Unresponsive/-Intolerant High-Risk Non-Muscle-Invasive Bladder Cancer: An Open-Label, Randomized, Multicenter, Phase 2 Study
Brief Title: Toripalimab ± Sequential Intravesical Gemcitabine-Mitomycin C for BCG-Unresponsive/-Intolerant High-Risk NMIBC: Open-Label Randomized Phase 2 Study
Acronym: OHAI-NMIBC-01
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: First Affiliated Hospital of Wenzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KY2025-352
Record Dates: First submitted 2025-09-17; First posted 2025-09-24 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Urinary Bladder Neoplasms; Carcinoma, Transitional Cell; Carcinoma in Situ of Bladder; Non-Muscle-Invasive Bladder Cancer
Keywords: NMIBC; High-Risk NMIBC; BCG-Unresponsive; BCG-Intolerant; BCG Failure; Carcinoma in Situ (CIS); Intravesical Therapy; Ta; T1; Gemcitabine; Mitomycin C; GEM-MMC; Toripalimab; PD-1 Inhibitor; Bladder-Sparing
MeSH Terms: conditions — Urinary Bladder Neoplasms; Carcinoma, Transitional Cell; Non-Muscle Invasive Bladder Neoplasms; Carcinoma in Situ | interventions — toripalimab; Gemcitabine; Mitomycin

STUDY DESIGN:
Intervention Model Description: Two-arm, 1:1 randomised, open-label, parallel-group phase 2 trial comparing toripalimab plus sequential intravesical gemcitabine→mitomycin C with toripalimab alone in adults with BCG-unresponsive or BCG-intolerant high-risk NMIBC. Randomisation stratified by CIS status, stage (Ta vs T1), BCG failure subtype, and study centre. Treatment up to 24 months.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Combination: Toripalimab + Intravesical GEM-MMC (Experimental): Toripalimab IV Q3W starting with the first intravesical cycle, plus sequential intravesical gemcitabine followed by mitomycin C in the same visit. Induction weekly ×6; if no recurrence at first tumour assessment (~month 3), monthly maintenance up to 24 months.
  Interventions: Drug: Toripalimab; Drug: Gemcitabine (GEM); Drug: Mitomycin C (MMC)
- Monotherapy: Toripalimab Alone (Active Comparator): Toripalimab IV every 3 weeks (Q3W) up to 24 months or until disease progression, unacceptable toxicity, or withdrawal; no intravesical chemotherapy.
  Interventions: Drug: Toripalimab

INTERVENTIONS:
Drug: Toripalimab — PD-1 inhibitor administered intravenously every 3 weeks (Q3W) for up to 24 months. Starts during the first intravesical treatment cycle.
  Other Names: JS001; Tuoyi
Drug: Gemcitabine (GEM) — Intravesical instillation as part of a sequential regimen with mitomycin C: weekly for 6 weeks (induction); if no recurrence at first tumour assessment (~month 3), maintenance instillations continue monthly up to 24 months.
  Other Names: GEM
  Arms: Combination: Toripalimab + Intravesical GEM-MMC
Drug: Mitomycin C (MMC) — Intravesical instillation immediately after intravesical gemcitabine in the same visit (sequential regimen): weekly for 6 weeks (induction); if eligible, monthly maintenance up to 24 months.
  Arms: Combination: Toripalimab + Intravesical GEM-MMC

SUMMARY:
This open-label, randomised, multicentre, phase 2 study (OHAI-NMIBC-01) compares toripalimab plus sequential intravesical gemcitabine followed by mitomycin C (GEM→MMC) with toripalimab alone in adults with BCG-unresponsive or BCG-intolerant high-risk non-muscle-invasive bladder cancer (HR-NMIBC). Two prespecified cohorts are analysed: (1) CIS cohort (CIS with/without Ta/T1) and (2) non-CIS cohort (high-risk Ta/T1 without CIS). In the combination arm, intravesical GEM→MMC is given weekly for 6 weeks (induction) and, for patients without recurrence at the first tumour assessment (~month 3), monthly maintenance continues up to 24 months or until progression/unacceptable toxicity; toripalimab IV every 3 weeks starts during the first intravesical cycle and continues up to 24 months or until progression/unacceptable toxicity. The monotherapy arm receives toripalimab IV every 3 weeks up to 24 months or until progression/unacceptable toxicity. Cystoscopy and urine cytology are performed every 3 months; imaging every 24 weeks. Primary endpoints are 3-month complete response (CR) rate in the CIS cohort and median recurrence-free survival (RFS) in the non-CIS cohort. Secondary endpoints include landmark CR, PFS and OS, RFS/HG-RFS landmarks in the non-CIS cohort, and safety (CTCAE v5.0). Exploratory analyses will assess outcomes by protocol-defined PD-L1 status. Approximately 106 participants will be enrolled at multiple sites in China.

DETAILED DESCRIPTION:
Rationale and Objectives. A substantial proportion of HR-NMIBC patients are BCG-unresponsive or BCG-intolerant and face early high-grade recurrence and consideration of cystectomy. This trial evaluates whether adding sequential intravesical chemotherapy (gemcitabine followed by mitomycin C in the same visit) to systemic PD-1 blockade (toripalimab) improves outcomes versus toripalimab alone.

Design. Prospective, open-label, randomised (1:1), parallel-group, phase 2 study at multiple centres in China. Treatment continues until recurrence/progression, unacceptable toxicity, withdrawal, or completion of 24 months.

Interventions.

Arm A (Combination): Toripalimab 240 mg IV every 3 weeks (Q3W) up to 24 months plus intravesical GEM→MMC: gemcitabine 1,000 mg retained ~60 min and drained, then mitomycin C 40 mg retained ~60 min; administered weekly for 6 weeks (induction) and then maintenance every 4 weeks (Q4W) up to month 24 if no high-grade recurrence.

Arm B (Monotherapy): Toripalimab 240 mg IV Q3W up to 24 months.

Assessments. Cystoscopy and urine cytology at months 3, 6, 9, 12 and every 3 months thereafter; abdominopelvic/upper-tract CT or MRI every 24 weeks; routine laboratory tests prior to dosing/instillation. (Exploratory tissue/urine/blood sampling may be performed per protocol.)

Primary Endpoints.

CIS cohort: CR rate at month 3 (proportion). CR is met by any of the following protocol-specified scenarios indicating no high-grade bladder disease: (a) negative urine cytology and negative cystoscopy; (b) negative cytology with cystoscopic lesions that are benign or low-grade Ta on biopsy; or (c) negative cystoscopy with positive cytology attributed to tumour in the upper tract or prostatic urethra and random bladder biopsies negative.

Non-CIS cohort: Median RFS, defined as time from start of treatment to high-grade Ta recurrence, any T1, or new CIS. Recurrence requires cystoscopic suspicion confirmed by histopathology; if cytology becomes positive prior to histologic confirmation, the recurrence date is set at the first positive cytology once recurrence is subsequently confirmed.

Secondary Endpoints.

CIS cohort: CR rates at months 6, 12, 18, and 24; PFS rates at the same landmarks (progression defined as lamina propria invasion from Ta/CIS to T1, progression to ≥T2, or new nodal/distant metastasis); OS at month 24, EOT+6 months, and EOT+12 months; incidence of adverse events (AEs).

Non-CIS cohort: RFS rates at months 6, 12, 18, and 24; high-grade RFS (HG-RFS) rates at the same landmarks (high-grade recurrence defined as Tis or Ta/T1 high-grade, or muscle-invasive disease at TURBT or cystectomy); PFS rates at months 6/12/18/24; OS at month 24, EOT+6 months, and EOT+12 months; AE incidence.

Exploratory Endpoints.

CIS cohort: 3-month CR rate in PD-L1-positive and PD-L1-negative subgroups (per protocol-specified assay and criteria; no prespecified CPS threshold).

Non-CIS cohort: Median RFS in PD-L1-positive and PD-L1-negative subgroups (recurrence definitions as above).

Sample Size and Oversight. Approximately 106 participants will be randomised 1:1. Safety will be monitored throughout; a Data Monitoring Committee oversees participant protection and study conduct.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years; sex: all; signed written informed consent by the participant or legally authorised representative.
2. Histologically confirmed high-risk non-muscle-invasive bladder cancer (HR-NMIBC), defined as any T1, high-grade Ta, and/or carcinoma in situ (CIS).
3. BCG-intolerant (unable to continue BCG because of severe adverse reactions) or meeting at least one definition of BCG treatment failure:

   1. Persistent or recurrent CIS within 12 months after completion of adequate BCG (with or without concomitant NMIBC);
   2. Recurrent high-grade Ta/T1 within 6 months after completion of adequate BCG;
   3. High-grade T1 at the first evaluation after BCG induction (~3 months);
   4. Ta high-grade and/or CIS present or recurrent at ~3 months after receiving ≥5 BCG instillations.

   Adequate BCG, for the purposes of this protocol, is defined as receipt of at least 5 of 6 induction instillations (maintenance not required).
4. ECOG performance status 0-2.
5. Adequate organ function per protocol laboratory criteria.
6. No intravesical chemotherapy or immunotherapy between the most recent cystoscopy/TURBT and study start; a single immediate postoperative intravesical chemotherapy at the time of the most recent cystoscopy/TURBT is allowed during screening per local practice.
7. Willing and able to comply with study procedures.

Exclusion Criteria:

1. Muscle-invasive bladder cancer (T2-T4).
2. Low-grade (LG) recurrence during or after BCG therapy.
3. Concomitant upper tract urothelial carcinoma, or lymph-node/distant metastasis.
4. Indwelling ureteral stent or known vesicoureteral reflux.
5. Contraindications to intravesical instillation, including within 2 weeks after TURBT, bladder perforation, symptomatic urinary tract infection, or gross haematuria.
6. Known hypersensitivity or contraindication to gemcitabine, mitomycin C, or toripalimab.
7. Systemic chemotherapy, small-molecule targeted therapy, or radiotherapy within 2 weeks before first study treatment.
8. Prior immune checkpoint inhibitor therapy.
9. Pregnant, planning pregnancy, or breastfeeding women.
10. Ongoing acute or chronic systemic infection, or history of active tuberculosis.
11. Other malignancy requiring active treatment.
12. Any condition that, in the investigator's judgment, makes participation not in the patient's best interest or could confound study results.

Study Population Adults with BCG-unresponsive or BCG-intolerant HR-NMIBC treated at participating centres in China.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2027-10 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
Complete Response (CR) Rate at Month 3 in the CIS Cohort | Baseline to Month 3
  Proportion of participants in the CIS cohort achieving CR at month 3. CR is met by any of the following protocol-specified scenarios indicating no high-grade bladder disease: (a) negative urine cytology and negative cystoscopy; (b) negative cytology with cystoscopic lesions that are benign or low-grade Ta on biopsy; or (c) negative cystoscopy with positive cytology attributed to tumour in the upper tract or prostatic urethra and random bladder biopsies negative.
Median Recurrence-Free Survival (RFS) in the Non-CIS Cohort | From randomisation/start of treatment to first event, assessed up to 24 months
  RFS is time to high-grade Ta recurrence, any T1, or new CIS, whichever occurs first. Recurrence requires cystoscopic suspicion confirmed by histopathology; if cytology becomes positive before histologic confirmation, the recurrence date is set at the first positive cytology once recurrence is subsequently confirmed. Death from any cause before documented recurrence is counted as an event.

SECONDARY OUTCOMES:
CR Rates at Months 6, 12, 18, and 24 in the CIS Cohort | Baseline to months 6, 12, 18, and 24
  Proportion of participants in the CIS cohort with CR at the specified time points using the protocol CR definition.
Progression-Free Survival (PFS) Rates at Months 6, 12, 18, and 24 in the CIS Cohort | Baseline to months 6, 12, 18, and 24
  Proportion without progression at each time point. Progression is defined as lamina propria invasion from Ta/CIS to T1, or progression to ≥T2, or new nodal or distant metastasis.
Overall Survival at Month 24, EOT+6 Months, and EOT+12 Months in the CIS Cohort | Baseline to Month 24, EOT+6 months, and EOT+12 months
  Survival status at prespecified landmarks.
Incidence of Adverse Events in the CIS Cohort | From first dose/instillation to 90 days post-last dose/instillation (≈ up to 27 months)
  Participants with treatment-emergent AEs and grade ≥3 AEs (MedDRA; CTCAE v5.0). Immune-related and instillation-related events summarised.
Recurrence-Free Survival Rates at Months 6, 12, 18, and 24 in the Non-CIS Cohort | Baseline to months 6, 12, 18, and 24
  Proportion without recurrence (high-grade Ta, any T1, or new CIS) or death at each time point; recurrence confirmation rules per protocol.
High-Grade Recurrence-Free Survival (HG-RFS) Rates at Months 6, 12, 18, and 24 in the Non-CIS Cohort | Baseline to months 6, 12, 18, and 24
  Proportion without high-grade recurrence at each time point. High-grade recurrence is defined as Tis or Ta/T1 high-grade, or muscle-invasive disease identified at TURBT or cystectomy.
Progression-Free Survival Rates at Months 6, 12, 18, and 24 in the Non-CIS Cohort | Baseline to Months 6, 12, 18, and 24
  Proportion without progression (lamina propria invasion from Ta/CIS to T1, progression to ≥T2, or new nodal/distant metastasis). Death before documented progression counts as an event.
Overall Survival at Month 24, EOT+6 Months, and EOT+12 Months in the Non-CIS Cohort | Baseline to Month 24, EOT+6 months, and EOT+12 months
  Survival status at prespecified landmarks.
Incidence of Adverse Events in the Non-CIS Cohort | From first dose/instillation to 90 days post-last dose/instillation (≈ up to 27 months)
  Participants with treatment-emergent AEs and grade ≥3 AEs (MedDRA; CTCAE v5.0).

OTHER OUTCOMES:
CR Rate at Month 3 in PD-L1-Positive Participants in the CIS Cohort | Baseline to Month 3
  Proportion of PD-L1-positive participants in the CIS cohort who achieve CR at Month 3. CR is met by any of: (a) negative urine cytology and negative cystoscopy; (b) negative cytology with cystoscopic lesions that are benign or low-grade Ta on biopsy; or (c) negative cystoscopy with positive cytology attributed to tumour in the upper tract or prostatic urethra and random bladder biopsies negative.
CR Rate at Month 3 in PD-L1-Negative Participants in the CIS Cohort | Baseline to Month 3
  Proportion of PD-L1-negative participants in the CIS cohort who achieve CR at Month 3; CR definition as above.
Median Recurrence-Free Survival in PD-L1-Positive Participants in the Non-CIS Cohort | From randomisation/start of treatment to first event, up to 24 months
  RFS is time from randomisation/start of treatment to high-grade Ta recurrence, any T1, or new CIS, whichever occurs first. Recurrence requires cystoscopic suspicion confirmed by histopathology; if cytology becomes positive before histologic confirmation, the event date is the first positive cytology once recurrence is subsequently confirmed. Death before recurrence counts as an event.
Median Recurrence-Free Survival in PD-L1-Negative Participants in the Non-CIS Cohort | From randomisation/start of treatment to first event, up to 24 months
  RFS definition and event-dating rules as above.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided
The sponsor and investigators intend to share de-identified IPD but the final plan (scope, timing, and access mechanism) is pending institutional approvals. This record will be updated once the IPD sharing policy is finalised.

REFERENCES:
- [Background] Holzbeierlein JM, Bixler BR, Buckley DI, Chang SS, Holmes R, James AC, Kirkby E, McKiernan JM, Schuckman AK. Diagnosis and Treatment of Non-Muscle Invasive Bladder Cancer: AUA/SUO Guideline: 2024 Amendment. J Urol. 2024 Apr;211(4):533-538. doi: 10.1097/JU.0000000000003846. Epub 2024 Jan 24. PMID 38265030
- [Background] Lightfoot AJ, Breyer BN, Rosevear HM, Erickson BA, Konety BR, O'Donnell MA. Multi-institutional analysis of sequential intravesical gemcitabine and mitomycin C chemotherapy for non-muscle invasive bladder cancer. Urol Oncol. 2014 Jan;32(1):35.e15-9. doi: 10.1016/j.urolonc.2013.01.009. Epub 2013 Mar 17. PMID 23510863
- [Background] Breyer BN, Whitson JM, Carroll PR, Konety BR. Sequential intravesical gemcitabine and mitomycin C chemotherapy regimen in patients with non-muscle invasive bladder cancer. Urol Oncol. 2010 Sep-Oct;28(5):510-4. doi: 10.1016/j.urolonc.2008.11.019. Epub 2009 Jan 26. PMID 19171491
- [Background] Black PC, Tangen CM, Singh P, McConkey DJ, Lucia MS, Lowrance WT, Koshkin VS, Stratton KL, Bivalacqua TJ, Kassouf W, Porten SP, Bangs R, Plets M, Thompson IM Jr, Lerner SP. Phase 2 Trial of Atezolizumab in Bacillus Calmette-Guerin-unresponsive High-risk Non-muscle-invasive Bladder Cancer: SWOG S1605. Eur Urol. 2023 Dec;84(6):536-544. doi: 10.1016/j.eururo.2023.08.004. Epub 2023 Aug 16. PMID 37596191
- [Background] Necchi A, Roumiguie M, Kamat AM, Shore ND, Boormans JL, Esen AA, Lebret T, Kandori S, Bajorin DF, Krieger LEM, Niglio SA, Uchio EM, Seo HK, de Wit R, Singer EA, Grivas P, Nishiyama H, Li H, Baranwal P, Van den Sigtenhorst-Fijlstra M, Kapadia E, Kulkarni GS. Pembrolizumab monotherapy for high-risk non-muscle-invasive bladder cancer without carcinoma in situ and unresponsive to BCG (KEYNOTE-057): a single-arm, multicentre, phase 2 trial. Lancet Oncol. 2024 Jun;25(6):720-730. doi: 10.1016/S1470-2045(24)00178-5. Epub 2024 May 10. PMID 38740030
- [Background] Balar AV, Kamat AM, Kulkarni GS, Uchio EM, Boormans JL, Roumiguie M, Krieger LEM, Singer EA, Bajorin DF, Grivas P, Seo HK, Nishiyama H, Konety BR, Li H, Nam K, Kapadia E, Frenkl T, de Wit R. Pembrolizumab monotherapy for the treatment of high-risk non-muscle-invasive bladder cancer unresponsive to BCG (KEYNOTE-057): an open-label, single-arm, multicentre, phase 2 study. Lancet Oncol. 2021 Jul;22(7):919-930. doi: 10.1016/S1470-2045(21)00147-9. Epub 2021 May 26. PMID 34051177
- See also: EAU Guidelines on Non-muscle-invasive Bladder Cancer (TaT1 and CIS) — https://uroweb.org/guidelines/non-muscle-invasive-bladder-cancer